CLINICAL TRIAL: NCT01467115
Title: Induction Chemotherapy With Taxotere, Cisplatin and 5-Fluorouracil Followed by Concomitant Cetuximab and Radiation for Locoregionally Advanced Squamous Cell Cancer of the Head and Neck: A Phase II Trial
Brief Title: Induction Chemotherapy Followed by Cetuximab and Radiation Therapy for Head and Neck Cancer
Acronym: DREXNECK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19834
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: loco regionally advanced; head and neck cancer; chemotherapy; radiation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Leucovorin; Cetuximab; Filgrastim; Erythropoietin; Epoetin Alfa; Cisplatin; Fluorouracil; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment with induction chemotherapy followed by radiation and cetuximab.
  Interventions: Radiation: Radiotherapy; Drug: Leucovorin; Biological: Cetuximab; Drug: Filgrastim; Drug: Erythropoetin; Drug: Cisplatin; Drug: Fluorouracil; Drug: Docetaxel

INTERVENTIONS:
Radiation: Radiotherapy — 3D conformal radiation therapy or Intensity-Modulated Radiation Therapy (IMRT) with or without Image Guided Radiation Therapy (IGRT) will be used for all patients. Radiotherapy will be delivered in 1.8 to 2.25 Gy fractions daily, five days per week excluding holidays, for a total of 66-72 Gy delivered to the Gross Tumor Volume (GTV, defined below) plus appropriate margin and 44-59.4 Gy to at-risk lymph nodes as determined by primary tumor characteristics. Alternative fractionation and dosing schema may be used as deemed appropriate for an individual case. For IMRT, the minimum Planning Target Volume (PTV) dose should be 90% of the prescription dose and a minimum of 95% of the PTV should receive the prescribed dose.
  Other Names: 3D conformal radiation therapy; Intensity-Modulated Radiation Therapy (IMRT)
Drug: Leucovorin — 5FU is given after, or at the midpoint, of the leucovorin infusion. Leucovorin is usually administered by I.V. bolus injection or short (10-120 minutes) I.V. infusion but oral formulation may be substituted should supply warrant.
  Other Names: Folinic acid, Leucovorin Ca.
Biological: Cetuximab — Cetuximab will be given for the duration of radiotherapy. A loading dose of intravenous cetuximab at 400mg per square meter body-surface area will be given over two hours up to seven days prior to initiation of radiation treatments or on the day of the first treatment (drug information detailed below). Thereafter, cetuximab will be given weekly over 60 minutes at a dose of 250 mg per meter squared. Intravenous diphenhydramine (50 mg) will be given as premedication.
  Other Names: Erbitux
Drug: Filgrastim — Neupogen®: 300 mcg/mL (1 mL, 1.6 mL). May be administered undiluted by SubQ injection. May also be administered by I.V. bolus over 15-30 minutes in D5W, or by continuous SubQ or I.V. infusion. Do not administer earlier than 24 hours after or in the 24 hours prior to cytotoxic chemotherapy.
  Other Names: Neupogen
Drug: Erythropoetin — Subcutaneous or intravenous
  Other Names: Epogen®; Procrit®
Drug: Cisplatin — One cycle of induction chemotherapy will be comprised of docetaxel on day 1 and cisplatin and 5-fluorouracil given days 1, 8, and 15. Intravenous docetaxel will be administered over one hour at a dose of 75 mg per square meter of body-surface area, followed by intravenous cisplatin at 35 mg per square meter, administered during a period of 0.5 to 3 hours weekly. After completion of the cisplatin infusion, intravenous fluorouracil will be given as a bolus at 1000 mg per square meter, followed by leucovorin at the dose of 350mg/m2. There will be total 4 cycles of chemotherapy of which 2 cycles will be prior to radiation therapy and 2 cycles will be post-radiation.
  Other Names: Platinol AQ
Drug: Fluorouracil — One cycle of induction chemotherapy will be comprised of docetaxel on day 1 and cisplatin and 5-fluorouracil given days 1, 8, and 15. Intravenous docetaxel will be administered over one hour at a dose of 75 mg per square meter of body-surface area, followed by intravenous cisplatin at 35 mg per square meter, administered during a period of 0.5 to 3 hours weekly. After completion of the cisplatin infusion, intravenous fluorouracil will be given as a bolus at 1000 mg per square meter, followed by leucovorin at the dose of 350mg/m2. There will be total 4 cycles of chemotherapy of which 2 cycles will be prior to radiation therapy and 2 cycles will be post-radiation.
Drug: Docetaxel — One cycle of induction chemotherapy will be comprised of docetaxel on day 1 and cisplatin and 5-fluorouracil given days 1, 8, and 15. Intravenous docetaxel will be administered over one hour at a dose of 75 mg per square meter of body-surface area, followed by intravenous cisplatin at 35 mg per square meter, administered during a period of 0.5 to 3 hours weekly. After completion of the cisplatin infusion, intravenous fluorouracil will be given as a bolus at 1000 mg per square meter, followed by leucovorin at the dose of 350mg/m2. There will be total 4 cycles of chemotherapy of which 2 cycles will be prior to radiation therapy and 2 cycles will be post-radiation.
  Other Names: Taxotere

SUMMARY:
More than 50% of Head and Neck cancers are locally advanced at presentation. Although surgery, in combination with other modalities like radiation therapy can achieve 40-50% five year survival rates, resection in the head and neck region can leave patients with poor functional and cosmetic outcomes.

Due to these concerns about quality of life after surgery, there has been a lot of interest in non surgical alternatives of treatment. Various combinations of radiation, chemotherapy and biologics has showed promising results. However, questions still remain about the ideal combination treatment regimen.

Based on assimilation of data from multiple sources, our study tries to identify the role of a potentially highly effective multi-modality regimen based on induction chemotherapy (Cisplatin, Docetaxel and 5 Fluorouracil) followed by combination of a biologic agent, Cetuximab, and radiation therapy.

DETAILED DESCRIPTION:
Patients will be given two cycles of induction chemotherapy with Cisplatin, Docetaxel and Fluorouracil. This will be followed by six weeks of radiation therapy along with Cetuximab. Patients will get two more cycles of chemotherapy with the same agents after the completion of radiation therapy course. Patients will be watched very closely during the trial period, with close follow up of treatment responses and monitoring of any adverse effects.

ELIGIBILITY:
INCLUSION CRITERIA

* Biopsy and/or fine needle aspirate of the tumor is required prior to registration. Pathologically confirmed primary squamous cell cancer of the oral cavity, oropharynx, hypopharynx, larynx, or unknown primary confined to the head and neck; histological variants such as spindle cell carcinoma, poorly differentiated keratin-positive carcinoma, and lymphoepithelioma are included. Patients with nasopharyngeal and salivary gland tumors are ineligible.
* Measureable disease representing stage III or stage IVa or IVb cancer by AJCC staging is required (See Appendix II)
* Measureable disease representing stage II cancer qualifies if the patient refuses surgery or is unable to undergo surgery as curative treatment
* Patient must not have had previous irradiation or surgery other than biopsy of the head and neck region
* A CT of the chest and CT or MRI of the tumor site is required within four weeks prior to registration
* Appropriate staging evaluation is required within four weeks prior to registration, including the following:
* history and physical examination with special attention to functional status measures, carotid arteries, neck and clavicular lymph nodes
* chest CT with evaluation of any nodules ≥ 1cm with biopsy or PET/CT (patients with lesions < 1cm, negative on PET scan, or that cannot be safely biopsied remain eligible).
* ECOG performance status 0-2 (See Appendix III)
* Age ≥ 18 years
* Complete blood count evaluation within two weeks of treatment demonstrating absolute neutrophil count ≥ 1500/mm3, platelets ≥100,000 cells/mm3, and hemoglobin ≥ 8g/dL
* Liver function tests within two weeks of treatment demonstrating total bilirubin ≤1.5 mg/dL, AST and ALT < 2x upper limit of normal, and alkaline phosphatase < 2x upper limits of normal; an abdominal CT scan is required if any of the above criteria are not met
* Adequate renal function measured within two weeks of treatment, defined as a creatinine clearance ≥ 50 ml/min determined by a 24 hour urine creatinine or the Cockcroft-Gault equation, where creatinine clearance (ml/min) is equal to:

[(140 - age) x (wt in kg)] x 0.85 for females [(sCR) x (72)]

* Corrected serum calcium <11 mg/dL within two weeks prior to treatment.
* Urine pregnancy test two weeks prior to treatment for women of childbearing potential; women of childbearing potential and male participants must agree to use a medically effective means of contraception throughout the duration of treatment and 30 days thereafter
* All patients must sign study-specific informed consent prior to study entry.

EXCLUSION CRITERIA:

* Evidence of metastatic disease
* Prior head and neck cancer.
* History of invasive cancer of any primary sight not considered cured.
* Previous radiation to the head and neck
* Nasopharyngeal or salivary gland cancer
* Severe, active comorbidity, defined as:
* New York Heart Association Class III or IV heart failure (Appendix IV)
* Unstable angina
* Acute bacterial or fungal infection requiring antibiotic treatment
* Chronic obstructive pulmonary disease requiring long term oral steroids or hospitalization for exacerbation within three months of study registration
* Liver dysfunction resulting in clinical jaundice or coagulation defects
* Acquired Immune Deficiency Syndrome defined as CD4 count <200 or opportunistic AIDS defining infection requiring active antibiotic treatment
* Pregnancy, lactation, or refusal of patient to take appropriate medical or behavioral measures to prevent pregnancy
* Pre-existing peripheral neuropathy > grade 2
* Hypersensitivity reaction to any drug listed in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-03; Primary Completion 2014-06 (Actual); Study Completion 2014-10-07 (Actual)

PRIMARY OUTCOMES:
Organ Sparing Survival | 3 years
  to determine whether the intervention will prolong survival without needing salvage surgery (organ sparing survival)

SECONDARY OUTCOMES:
Overall Survival | 3 years
  we will determine if the intervention prolongs overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Rene R Rubin, MD, Principal Investigator — Drexel University
Locations (1):
- Hahnemann University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haddad RI, Shin DM. Recent advances in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1143-54. doi: 10.1056/NEJMra0707975. No abstract available. PMID 18784104
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Deshmane VH, Parikh HK, Pinni S, Parikh DM, Rao RS. Laryngectomy: a quality of life assessment. Indian J Cancer. 1995 Sep;32(3):121-30. PMID 8772812
- [Background] De Boer MF, McCormick LK, Pruyn JF, Ryckman RM, van den Borne BW. Physical and psychosocial correlates of head and neck cancer: a review of the literature. Otolaryngol Head Neck Surg. 1999 Mar;120(3):427-36. doi: 10.1016/S0194-5998(99)70287-1. PMID 10064650
- [Background] Department of Veterans Affairs Laryngeal Cancer Study Group; Wolf GT, Fisher SG, Hong WK, Hillman R, Spaulding M, Laramore GE, Endicott JW, McClatchey K, Henderson WG. Induction chemotherapy plus radiation compared with surgery plus radiation in patients with advanced laryngeal cancer. N Engl J Med. 1991 Jun 13;324(24):1685-90. doi: 10.1056/NEJM199106133242402. PMID 2034244
- [Background] Paccagnella A, Orlando A, Marchiori C, Zorat PL, Cavaniglia G, Sileni VC, Jirillo A, Tomio L, Fila G, Fede A, et al. Phase III trial of initial chemotherapy in stage III or IV head and neck cancers: a study by the Gruppo di Studio sui Tumori della Testa e del Collo. J Natl Cancer Inst. 1994 Feb 16;86(4):265-72. doi: 10.1093/jnci/86.4.265. PMID 8158680
- [Background] Zorat PL, Paccagnella A, Cavaniglia G, Loreggian L, Gava A, Mione CA, Boldrin F, Marchiori C, Lunghi F, Fede A, Bordin A, Da Mosto MC, Sileni VC, Orlando A, Jirillo A, Tomio L, Pappagallo GL, Ghi MG. Randomized phase III trial of neoadjuvant chemotherapy in head and neck cancer: 10-year follow-up. J Natl Cancer Inst. 2004 Nov 17;96(22):1714-7. doi: 10.1093/jnci/djh306. PMID 15547184
- [Background] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544